CLINICAL TRIAL: NCT07188649
Title: Early Postoperative SpO₂/FiO₂ Ratio in Obese and Non-Obese Patients Undergoing Laparoscopic Surgery in the Reverse Trendelenburg Position: Evaluation Together With the STOP-BANG Score
Brief Title: Postoperative SpO₂/FiO₂ in Obese and Non-Obese Patients: Role of STOP-BANG
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, Assoc. prof, Haseki Training and Research Hospital
Other Study IDs: hulusi tez
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Oxygen Deficiency
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- obese: BMI ≥ 35
  Interventions: Behavioral: oxygen deficiency
- control: BMI < 35
  Interventions: Behavioral: oxygen deficiency

INTERVENTIONS:
Behavioral: oxygen deficiency — The aim of this study is to evaluate the effect of the Reverse Trendelenburg position on oxygenation (SpO₂/FiO₂ ratio) in the early postoperative period in patients undergoing laparoscopic surgery. In our study, obesity is considered as a comparative subgroup in terms of variability of this effect; additionally, the STOP-BANG score, which measures the risk of obstructive sleep apnea syndrome, is examined as an auxiliary indicator.

SUMMARY:
The aim of this study is to evaluate the effect of the Reverse Trendelenburg position on oxygenation (SpO₂/FiO₂ ratio) in the early postoperative period in patients undergoing laparoscopic surgery. In our study, obesity is considered as a comparative subgroup in terms of variability of this effect; additionally, the STOP-BANG score, which measures the risk of obstructive sleep apnea syndrome, is examined as an auxiliary indicator.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patients who give consent to participate in the study
* Patients who underwent elective laparoscopic cholecystectomy in Reverse Trendelenburg (30 degrees) position
* ASA I-III patients
* Patients with operation time < 3 hours

Exclusion Criteria:

* Patients under 18 years old
* Patients who did not give consent
* Patients with asthma, COPD, or known respiratory disease
* Patients whose procedure could not be completed or who had missing data
* Patients with general anesthesia duration < 90 minutes will not be included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults over 18, ASA I-III patients, patients who give consent to participate, patients undergoing elective laparoscopic surgery (obesity surgery, cholecystectomy, umbilical hernia, etc.)
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
oxygen level | 4 months
  SpO₂/FiO₂ ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Üniversity, Istanbul, Merkez Mahallesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Michael Dunham C, Hileman BM, Hutchinson AE, Antonaccio T, Chance EA, Huang GS, Szmaj G, Calabro K, Bishop C, Schrickel TT. Evaluation of operating room reverse Trendelenburg positioning and its effect on postoperative hypoxemia, aspiration, and length of stay: a retrospective study of consecutive patients. Perioper Med (Lond). 2017 Aug 22;6:10. doi: 10.1186/s13741-017-0067-2. eCollection 2017. PMID 28852473
- [Result] 5. Pirenne S, Hans G, Leloup von Edelsberg S, Joris J. STOP-BANG but not BMI predicts postoperative obstructive apnea and hypoxemia after laparoscopic upper-abdominal surgery. University of Liège, Department of Anaesthesiology & Intensive Care, Belgium.